CLINICAL TRIAL: NCT02131389
Title: Non-Randomized, Multi-Site, Post-Market Study of the ICONACY I-Hip System (Protocol No. PS-1001)
Brief Title: Multi-Site, Post-Market Study of the ICONACY I-Hip System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iconacy Orthopedic Implants, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PS-1001
Record Dates: First submitted 2014-04-28; First posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Degenerative Joint Disease
Keywords: Hip; Arthroplasty; Arthroplasties; Prosthesis; Iconacy; Osteoarthritis; Arthritis; THA; THR; DJD
MeSH Terms: conditions — Joint Diseases; Osteoarthritis; Arthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Iconacy Hip System (Other): Iconacy hip system prosthesis components
  Interventions: Device: Iconacy Hip System

INTERVENTIONS:
Device: Iconacy Hip System
  Other Names: Iconacy I-Hip; I-Hip; iHip

SUMMARY:
The purpose of this study is to evaluate the use and efficacy of the I-Hip for primary total hip replacement surgery.

ELIGIBILITY:
Inclusion Criteria:

* A candidate for primary hip replacement on this operative hip.
* Is 30 to 80 years of age.
* Has hip joint disease related to one or more of the following:

  * Degenerative joint disease, (including osteoarthritis or post-traumatic arthritis)
  * Avascular Necrosis (AVN).
* Will be available for evaluation for the duration of the study.
* Is able and willing to speak and read English, read and sign the informed consent, fill out the WOMAC and Patient Satisfaction questionnaires, and follow all study procedures.

Exclusion Criteria:

* Is younger than 30 years of age or older than 80 years of age.
* Has undergone partial hip replacement or previous ORIF (open reduction internal fixation of femur or acetabulum).
* Has undergone total hip replacement on this hip in the past (no revisions allowed in study).
* Infection, or history of infection, acute or chronic, in the hip joint, or acute or chronic unresolved systemic infection.
* Is currently experiencing radicular pain from the spine down operative leg.
* Has participated in an IDE/IND clinical investigation with an investigational product in the last three months, or is involved in any personal injury litigation, medical-legal or worker's compensation claim.
* Is a known drug or alcohol abuser or has a psychological disorder that could affect the ability to complete patient reported questionnaires.
* Has been diagnosed with fibromyalgia or has a significant neurological or musculoskeletal disorder or disease that may adversely affect gait or weight bearing (e.g. muscular dystrophy, multiple sclerosis, Charcot disease).
* Has been diagnosed with Paget's disease or Congenital hip deformity (dysplasia and/or dislocation).
* Is suffering from inflammatory arthritis (e.g. rheumatoid arthritis, juvenile rheumatoid arthritis, psoriatic arthritis, systemic lupus erythematosus, etc.)
* Is Obese: (Defined for this study as having a BMI>45).
* Has insufficient bone quality.
* Has loss of ligamentous structures.
* Has materials sensitivity.
* Is currently a prisoner.
* Is pregnant or lactating.
* Has a contralateral amputation.
* Has a medical condition with less than 2 years of life expectancy.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2014-04; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic Success as a Measure of Radiolucency and Component Migration | 2 years
  A subject will be considered a failure for Overall Radiographic Success if one or more of the below conditions are met:
  The subject will be considered a RADIOGRAPHIC FAILURE if:
  1. there is a complete radiolucent line> 3mm wide at the bone/cement interface or
  2. there is a >5 degree migration (shift) of the component or
  3. there is a >5 mm migration (shift) of the component.
Improvement of Harris Hip Score (with Charnley Score and other comorbidities considered) | 2 years
Patient satisfaction clinical assessment utilizing questionnaire | 2 years
  Clinical assessment of patient satisfaction will be made by utilizing a Patient Satisfaction (PS) questionnaire.

SECONDARY OUTCOMES:
Revision of Implant Prosthesis as a Measure of Efficacy | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Donald L Pomeroy, MD, Principal Investigator — Pomeroy & Rhoads Orthopaedics, Inc.
Locations (2):
- United States (2):
  - Baptist Health Louisville, Louisville, Kentucky
  - Sts. Mary & Elizabeth Hospital - KentuckyOne Health, Louisville, Kentucky